CLINICAL TRIAL: NCT01239966
Title: Safety and Efficacy of Combined Extracorporeal CO2 Removal and Renal Replacement Therapy in Patients With the Acute Respiratory Distress Syndrome and Acute Renal Failure
Brief Title: Pulmonary And Renal Support During Acute Respiratory Distress Syndrome
Acronym: PARSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, MD, MSc, Hôpital Européen Marseille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-A00397-32
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Renal Failure
Keywords: Acute Respiratory Distress syndrome; Acute renal Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Combined ECCOR and RRT — Insertion of a membrane oxygenator (Hilite 2400 LT, Medos, Germany) within an hemofilter circuit (M150,PrismaFlex, Hospal); either upstream or downstream of the hemofilter.

SUMMARY:
In patients presenting with the acute respiratory distress syndrome (ARDS), mechanical ventilation with low tidal volume (6 ml/kg predicted body weight) is the current gold standard for supportive care. However, despite a relative low tidal volume, approximatively one third of patients will experienced tidal hyperinflation, a phenomenon known to induce pulmonary and systemic inflammatory response. A further reduction of the tidal volume to 4 ml/kg (PBW) will prevent pulmonary area from tidal hyperinflation. As a result, hypercarbia and respiratory acidosis are commonly observed with such very low tidal ventilation. Extra corporeal CO2 removal is one of a mean to normalize arterial CO2 tension.

Patients with ARDS also frequently develop acute renal failure which may required Renal Replacement Therapy. Some data suggests that starting early the RRT may favor outcome.

The investigators hypothesized that a strategy combining ECCOR and RRT early in the course of patients presenting ARDS and acute renal failure will allow the tidal volume to be further reduced, providing lung protection, while avoiding the arterial CO2 tension to be increased.

For this purpose, the investigators sought to evaluate the safety and efficacy of adding a membranel oxygenator within an hemofiltration circuit, either upstream or downstream of the hemofilter.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Distress Syndrome according to the AECC definition
* Acute Renal Failure according to the RIFLE definition

Exclusion Criteria:

* Age < 18 years
* PaO2/FiO2 < 100 with FIO2 = 1 and PEEP > 18 cmH2O
* DNR order or death expected within the next 3 days
* Intracranial haemorrhage or hypertension
* Heparin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Arterial carbon dioxide reduction | 20 min
  20 % reduction of arterial carbon dioxide tension after 20 min of combined ECCOR and RRT

SECONDARY OUTCOMES:
Gas transfer measurement | 20 min, H1, H6, H12, H24, H36, H48 and H72.
  Measurement of PO2 and PCO2 before and after the membrane oxygenation
Arterial blood gases | 20 min, H1, H6, H12, H24, H36, H48 and H72.
  Measurement of arterial blood gases
carbon dioxide elimination (VCO2) | 20 min, H1, H6, H12, H24, H36, H48 and H72.
  Measurement of carbon dioxide elimination rate at the ventilator and at the membrane oxygenator
Respiratory mechanics and hemodynamic parameters | 20 min, H1, H6, H12, H24, H36, H48 and H72.
  Measurement of respiratory mechanics and hemodynamic parameters
Safety monitoring | 20 min, H1, H6, H12, H24, H36, H48 and H72.
  Continuous measurement of the differential pressure across the oxygenator membrane and across the hemofilter.
  Assessment of catheter dysfunction, clotting or disruption of the extra-corporeal circuit, clotting of the oxygenator membrane or of the hemofilter.
  Assessment of patient's haemorragic or thrombotic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Allardet-Servent, MD, Principal Investigator — Hopital Ambroise Pare
Locations (2):
- France (2):
  - Hopital Paul Desbief, Marseille
  - Hopital Ambroise Pare, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Result] Terragni PP, Del Sorbo L, Mascia L, Urbino R, Martin EL, Birocco A, Faggiano C, Quintel M, Gattinoni L, Ranieri VM. Tidal volume lower than 6 ml/kg enhances lung protection: role of extracorporeal carbon dioxide removal. Anesthesiology. 2009 Oct;111(4):826-35. doi: 10.1097/ALN.0b013e3181b764d2. PMID 19741487
- See also: information related to hospitals and investigators involved — http://www.hopitaux-ambroisepare-desbief.com/